CLINICAL TRIAL: NCT04470934
Title: PMCF - Study on the Performance/Safety of SeQuent® Sirolimus-Coated Balloon (SCB, Investigational Device) in Patients With Coronary Artery Disease
Brief Title: SeQuent® SCB "All Comers" Post Market Clinical Follow-up (PMCF)
Acronym: SCORE
Status: Active, not recruiting | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1913
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Myocardial Ischaemia
Keywords: Coronary Artery Disease; Myocardial Ischemia; drug-coated balloon catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SeQuent® SCB drug-coated balloon catheter — treatment of coronary artery disease with SeQuent® SCB of "real world" de-novo and restenotic lesions in native coronary arteries and coronary bypass grafts

SUMMARY:
The aim of the study is to assess continued safety and efficacy of the SeQuent® SCB. The product under investigation will be used in routine clinical practice according to the latest European Society of Cardiology (ESC) guidelines and according to the Instructions for Use (IFU). Those data that are obtained in routine clinical use will be documented in the Case Report Form (CRF).

DETAILED DESCRIPTION:
The objective of the study is to assess the continued safety and efficacy of SeQuent® SCB for the treatment of "real world" de-novo and restenotic lesions in native coronary arteries and coronary bypass grafts. Study goals are based on non-inferiority for Drug-Coated Balloon (DCB) compared to Paclitaxel-Coated Balloon (PCB) and Dru-eluting Stents (DES) (historical data) with 80% power. Primary and secondary outcome variables are international accepted parameters in stent-trials, which sufficiently describe the efficacy and safety of the investigated device and allow clinical conclusions. Additional attention will be paid to those patients who received, by observation, a shortened dual antiplatelet therapy (DAPT).

The aim of the study is to assess the safety and efficacy of the SeQuent® SCB in the treatment of coronary artery disease with reference vessel diameters between ≥ 2 mm and ≤ 4 mm with suitable lesion lengths. There is no limitation of lesion lengths. In case the lesion is longer than 34 mm, more than one stent needs to be used.

ELIGIBILITY:
Inclusion Criteria:

* All common significant coronary lesions
* Target lesion length >34mm need to be covered with at least 2 devices
* Patients eligible for this study must be at least 18 years of age
* The patient must fulfil the standard recommendations for percutaneous coronary intervention (PCI), based on the last ESC recommendations within his/ her regular treatment or that the use of the product has already been decided within the regular planning of the patient's treatment

Exclusion Criteria:

* Intolerance to sirolimus
* Allergy to components of the coating
* Pregnancy and lactation
* Complete occlusion of the treatment vessel because of an unsuccessfully re-canalized
* Cardiogenic shock
* Risk of an intraluminal thrombus
* Hemorrhagic diathesis or another disorder such as gastro-intestinal ulceration or cerebral circulatory disorders which restrict the use of platelet aggregation inhibitor therapy and anti-coagulation therapy
* Surgery shortly after myocardial infarction with indications of thrombus or poor coronary flow behavior
* Severe allergy to contrast media
* Lesions which are untreatable with PCI or other interventional techniques
* Patients with an ejection fraction of < 30 %
* Vascular reference diameter < 2.00 mm
* Treatment of the left stem (first section of the left coronary artery)
* Indication for a bypass surgery
* Contraindication for whichever accompanying medication is necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-armed, prospective, international, multi-center, post-market study in patients with coronary artery disease and indication for PCI either due to anginal symptoms and a relevant stenotic coronary lesion during angiography or due to documented ischemia by non-invasive or invasive functional testing.
  All patients who undergo a target intervention with the SCB will be followed for 12 and 24 months after initial PCI.
Sampling Method: Non-Probability Sample
Enrollment: 1302 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | at 12 months
  Target Lesion Failure (TLF): defined as the composite rate of target vessel myocardial infarction (TV-MI) or ischemia-driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | at 24 months
  Target Lesion Failure (TLF): defined as the composite rate of target vessel myocardial infarction (TV-MI) or ischemia-driven target lesion revascularization (TLR).
ischemia driven target lesion revascularization (TLR) | at 12 months
ischemia driven target lesion revascularization (TLR) | at 24 months
all-cause death, cardiac death | at 12 months
all-cause death, cardiac death | at 24 months
all myocardial infarction (MI) and target vessel myocardial infarction (TV-MI) | at 12 months
all myocardial infarction (MI) and target vessel myocardial infarction (TV-MI) | at 24 months
major adverse coronary event (MACE) | at 12 months
  major adverse coronary event (MACE): defined as composite of cardiovascular death, myocardial infarction or ischemia-driven target lesion revascularization
major adverse coronary event (MACE) | at 24 months
  major adverse coronary event (MACE): defined as composite of cardiovascular death, myocardial infarction or ischemia-driven target lesion revascularization
Dual Antiplatelet Therapy (DAPT) compliance | at 4 weeks
Dual Antiplatelet Therapy (DAPT) compliance | at 3 months
Probable or definite stent-thrombosis of In-stent treated lesions | accumulated at 12 months
Probable or definite stent-thrombosis of In-stent treated lesions | accumulated at 24 months
Procedural success | immediately after procedure
  final diameter stenosis < 30 % without flow-limiting dissections
Bleeding complications according to the Bleeding Academic Research Consortium (BARC) | accumulated at 3 months
Bleeding complications according to the Bleeding Academic Research Consortium (BARC) | accumulated at 12 months
Bleeding complications according to the Bleeding Academic Research Consortium (BARC) | accumulated at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Otto, MD, Principal Investigator — Universitätsklinikum Jena - Klinik für Innere Medizin I
Locations (1):
- Universitätsklinikum Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otto S, Diaz VAJ, Weilenmann D, Cuculi F, Nuruddin AA, Leibundgut G, Alfonso F, Wan Ahmad WA, Pyxaras S, Rittger H, Steen P, Gaede L, Schulze C, Wohrle J, Rosenberg M, Waliszewski MW. Crystalline sirolimus-coated balloon (cSCB) angioplasty in an all-comers, patient population with stable and unstable coronary artery disease including chronic total occlusions: rationale, methodology and design of the SCORE trial. BMC Cardiovasc Disord. 2023 Mar 31;23(1):176. doi: 10.1186/s12872-023-03187-x. PMID 37003986